CLINICAL TRIAL: NCT04812340
Title: Effect of High-Intensity Circuit Training Versus Low-Intensity Interval Training on Functional Strength and Weight Efficacy in Overweight and Obese Young Females.
Brief Title: Effect of HICT and LIIT on Functional Strength and Weight Efficacy in Overweight and Obese Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00924 Huma Nayab
Record Dates: First submitted 2021-03-07; First posted 2021-03-23 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Overweight and Obesity
Keywords: female; Quality of life; overweight; obesity; Exercise
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity Circuit training (Active Comparator): Intervention will consist of 6 series with 3 minutes rest period between the series. The series will consist of burpees, skipping, 1 legged squats, leg levers, and push-ups. the exercise volume will be increased progressively over 8 weeks.
  Interventions: Other: High intensity circuit training
- Low intensity interval training (Active Comparator): the intervention will consist of 4 series of Low-intensity exercises with 3 minutes of rest. the series will comprise of jogging and walking. the Exercise volume will be increased gradually.
  Interventions: Other: Low intensity interval training

INTERVENTIONS:
Other: High intensity circuit training — 6 series with 3 minutes rest between the series. each series will consist of 30 seconds each of burpees, skipping, lunges, 1- legged squat, leg levers, and push-ups with 30 seconds rest in between. the volume of exercise will be increased progressively over a period of 8 weeks.
  Arms: High intensity Circuit training
Other: Low intensity interval training — 4 series with 3 minutes rest in between. each series will consist of 10 minutes of jogging and 5 minutes walking with 30 seconds recovery in between. the volume of exercise will be increased progressively over a period of 8 weeks.
  Arms: Low intensity interval training

SUMMARY:
This study is aimed at determining the effects of high-intensity circuit training versus low-intensity circuit training on functional strength and weight efficacy in overweight and obese females.

DETAILED DESCRIPTION:
A high-intensity circuit promotes muscle mass and as a result, potentially reduces the incidence of cardiovascular disease and reduces the risk of death in the young population. Low-intensity interval training increases muscle circulation and improving the uptake of oxygen. Both high-intensity circuit training and low-intensity interval training enhance body composition, quality of life, functional fitness and decrease body mass index. These trainings also motivate participants to continue their exercise. This study will help us determine whether high intensity or low-intensity training is more helpful in improving the functional strength and weight efficacy in overweight and obese females. As obesity is on the rise in modern society, our results will help improve the quality of life of obese and overweight females.

ELIGIBILITY:
Inclusion Criteria:

* Females with BMI >25 kg/m2.
* Females not engaged in routine exercise programs in last 6 months

Exclusion Criteria:

* Females who are using weight loss products.
* Females having uncontrolled diabetes, thyroid disease, arthritis, cardiac diseases, asthma, hypertension, and recent trauma would not be included in the study.
* Females who are pregnant would not be included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Overweight and obesity are very common in modern society among young females.
Enrollment: 34 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Functional Strength testing | 8th week
  changes from baseline functional strength testing consist of leg levers, push-ups, one-legged squats, and burpees which will be performed as many times as possible in one minute. All tests will be performed with 3 minutes recovery period in between. The number of repetitions for each test will be counted per minute. And this would be repeated at baseline as well as after 8 weeks.

SECONDARY OUTCOMES:
weight efficacy scale | 8th week
  changes from baseline Weight efficacy lifestyle questionnaire measures the confidence of the participants in their weight loss ability. It ranges from 0(no confidence) to 10(very confidence)[18]. Its reliability and validity are very high and it can be used in research, clinical and educational fields.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Ladies club Gujranwala club, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sand AS, Emaus N, Lian O. Overweight and obesity in young adult women: A matter of health or appearance? The Tromso study: Fit futures. Int J Qual Stud Health Well-being. 2015 Sep 22;10:29026. doi: 10.3402/qhw.v10.29026. eCollection 2015. PMID 26400463
- [Background] Paoli A, Pacelli QF, Moro T, Marcolin G, Neri M, Battaglia G, Sergi G, Bolzetta F, Bianco A. Effects of high-intensity circuit training, low-intensity circuit training and endurance training on blood pressure and lipoproteins in middle-aged overweight men. Lipids Health Dis. 2013 Sep 3;12:131. doi: 10.1186/1476-511X-12-131. PMID 24004639
- [Background] Seo YG, Noh HM, Kim SY. Weight loss effects of circuit training interventions: A systematic review and meta-analysis. Obes Rev. 2019 Nov;20(11):1642-1650. doi: 10.1111/obr.12911. Epub 2019 Jul 19. PMID 31322317
- [Background] Sydora BC, Turner C, Malley A, Davenport M, Yuksel N, Shandro T, Ross S. Can walking exercise programs improve health for women in menopause transition and postmenopausal? Findings from a scoping review. Menopause. 2020 Aug;27(8):952-963. doi: 10.1097/GME.0000000000001554. PMID 32404793
- [Background] Sperlich B, Wallmann-Sperlich B, Zinner C, Von Stauffenberg V, Losert H, Holmberg HC. Functional High-Intensity Circuit Training Improves Body Composition, Peak Oxygen Uptake, Strength, and Alters Certain Dimensions of Quality of Life in Overweight Women. Front Physiol. 2017 Apr 3;8:172. doi: 10.3389/fphys.2017.00172. eCollection 2017. PMID 28420999
- [Background] Mastrangelo MA, MacFarlane S, Woodrow K, Conway E, Klitz DD, Mauriello K, Miller-Scales A, Nieves-Ventimeglia L, Galantino ML. Effect of circuit training on menopausal symptoms and quality of life. Journal of Women's Health Physical Therapy. 2010 May 1;34(2):58-63.
- [Background] Marshall KD, Muller BN, Krenz M, Hanft LM, McDonald KS, Dellsperger KC, Emter CA. Heart failure with preserved ejection fraction: chronic low-intensity interval exercise training preserves myocardial O2 balance and diastolic function. J Appl Physiol (1985). 2013 Jan 1;114(1):131-47. doi: 10.1152/japplphysiol.01059.2012. Epub 2012 Oct 25. PMID 23104696
- [Background] Foster VL, Hume GJ, Byrnes WC, Dickinson AL, Chatfield SJ. Endurance training for elderly women: moderate vs low intensity. J Gerontol. 1989 Nov;44(6):M184-8. doi: 10.1093/geronj/44.6.m184. PMID 2809105
- [Background] de Oliveira MF, Caputo F, Corvino RB, Denadai BS. Short-term low-intensity blood flow restricted interval training improves both aerobic fitness and muscle strength. Scand J Med Sci Sports. 2016 Sep;26(9):1017-25. doi: 10.1111/sms.12540. Epub 2015 Sep 15. PMID 26369387
- [Background] Cardozo DC, DE Salles BF, Mannarino P, Vasconcelos APS, Miranda H, Willardson JM, Simao R. The Effect of Exercise Order in Circuit Training on Muscular Strength and Functional Fitness in Older Women. Int J Exerc Sci. 2019 May 1;12(4):657-665. doi: 10.70252/YAOI2219. eCollection 2019. PMID 31156754
- [Background] Preusser BA, Winningham ML, Clanton TL. High- vs low-intensity inspiratory muscle interval training in patients with COPD. Chest. 1994 Jul;106(1):110-7. doi: 10.1378/chest.106.1.110. PMID 8020255
- [Background] Gibala MJ. High-intensity interval training: a time-efficient strategy for health promotion? Curr Sports Med Rep. 2007 Jul;6(4):211-3. No abstract available. PMID 17617995
- [Background] Ballesta-Garcia I, Martinez-Gonzalez-Moro I, Rubio-Arias JA, Carrasco-Poyatos M. High-Intensity Interval Circuit Training Versus Moderate-Intensity Continuous Training on Functional Ability and Body Mass Index in Middle-Aged and Older Women: A Randomized Controlled Trial. Int J Environ Res Public Health. 2019 Oct 30;16(21):4205. doi: 10.3390/ijerph16214205. PMID 31671584
- [Background] Ballesta-Garcia I, Martinez-Gonzalez-Moro I, Ramos-Campo DJ, Carrasco-Poyatos M. High-Intensity Interval Circuit Training Versus Moderate-Intensity Continuous Training on Cardiorespiratory Fitness in Middle-Aged and Older Women: A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Mar 10;17(5):1805. doi: 10.3390/ijerph17051805. PMID 32164314
- [Background] Sperlich B, Hahn LS, Edel A, Behr T, Helmprobst J, Leppich R, Wallmann-Sperlich B, Holmberg HC. A 4-Week Intervention Involving Mobile-Based Daily 6-Minute Micro-Sessions of Functional High-Intensity Circuit Training Improves Strength and Quality of Life, but Not Cardio-Respiratory Fitness of Young Untrained Adults. Front Physiol. 2018 May 9;9:423. doi: 10.3389/fphys.2018.00423. eCollection 2018. PMID 29867519
- [Background] Ojeda ÁH, Maliqueo SG, Barahona-Fuentes G. Validity and reliability of the Muscular Fitness Test to evaluate body strength-resistance. Apunts Sports Medicine. 2020 Oct 1;55(208):128-36.
- [Background] Schulz BR, McDonald MJ. Weight loss self-efficacy and modelled behaviour: gaining competence through example. Canadian Journal of Counselling and Psychotherapy. 2011;45(1).
- [Background] Singh HK, Mun VL, Barua A, Ali SZ, Swee WC. Application and validation of the weight efficacy lifestyle (WEL) questionnaire among type 2 diabetes mellitus patients in Malaysia. Mal J Nutr. 2018;24(3):427-0.
- [Background] Navidian, A., Reliability and validity of the weight efficacy lifestyle questionnaire in overweight and obese individuals. International Journal of Behavioral Sciences, 2009. 3(3): p. 217-222.
- [Background] Kim JW, Ko YC, Seo TB, Kim YP. Effect of circuit training on body composition, physical fitness, and metabolic syndrome risk factors in obese female college students. J Exerc Rehabil. 2018 Jun 30;14(3):460-465. doi: 10.12965/jer.1836194.097. eCollection 2018 Jun. PMID 30018934